CLINICAL TRIAL: NCT02169258
Title: Prognostic Impact of ROUtine Coronary CathETerization in Low Extremity ArTEry Disease Undergoing Percutaneous Transluminal Angioplasty (PIROUETTE-PTA Study)
Brief Title: Routine Coronary Catheterization in Low Extremity Artery Disease Undergoing Percutaneous Transluminal Angioplasty
Acronym: PIROUETTEPTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Tainan Municipal Hospital (Other); E-DA Hospital (Other); Kaohsiung Medical University (Other); National Taiwan University Hospital (Other); Buddhist Tzu Chi General Hospital (Other); Far Eastern Memorial Hospital (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Ting-Hsing Chao, Associate Professor and Attending Physician, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-103-023
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Peripheral Artery Disease; Coronary Artery Disease
Keywords: coronary artery disease; peripheral artery disease; percutaneous transluminal angioplasty; coronary angiography; revascularization; gene polymorphisms; microRNAs
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Selective Strategy (Placebo Comparator): non-invasive evaluation of possible myocardial ischemia by using DSE or dTS followed by coronary angiography if the test is positive for ischemia
  Interventions: Procedure: Systemic Strategy
- Registry (No Intervention): Clinical decisions are reached by consensus of operators, patients and family as usual care
- Systemic Strategy (Active Comparator): Routine coronary angiography before PTA without a previous non-invasive stress test
  Interventions: Procedure: Systemic Strategy

INTERVENTIONS:
Procedure: Systemic Strategy — Significant CAD needing further revascularization is defined as patients who have luminal stenosis > 70% of the major epicardial vessels and bypass graft vessel or their major branches (> 50% for left main trunk or in-stent restenotic lesion) with reference vessel larger than 2.5 mm in diameter and moderate area of vulnerable myocardium for ischemia. Intermediate stenotic lesions should be determined if they are hemodynamic significant by fractional flow reserve (FFR) (<=0.8). The choice of revascularization procedure, either percutaneous coronary intervention or coronary artery bypass surgery, depends on operator's or cardiovascular team's suggestion and patient's decision.
  Other Names: Routine Coronary Angiography before PTA
  Arms: Selective Strategy; Systemic Strategy

SUMMARY:
1. The prevalence of significant and complex obstructive coronary artery disease (CAD) is high in patients who have low extremity artery disease (LEAD).
2. Long-term prognosis of LEAD undergoing percutaneous transluminal angioplasty (PTA) remains poor and CAD is an independent predictor of total mortality after PTA.
3. This prospective randomized controlled trial will evaluate the prognostic effects of routine versus selective coronary angiography before PTA for LEAD and elucidate the potential mechanism.

DETAILED DESCRIPTION:
1. participants

   1. eligible participants are randomly assigned to systemic strategy or selective strategy

      * participants allocated to systemic strategy will receive routine coronary angiography before PTA without a previous non-invasive stress test
      * subjects allocated to selective strategy will undergo non-invasive evaluation of possible myocardial ischemia by using dobutamine stress echocardiography (DSE) or dipyridamole thallium 201 myocardial perfusion scintigraphy (dTS) followed by coronary angiography if the test is positive for ischemia
   2. participants who are not willing to be randomized will be included in the registration group
2. revascularization

   1. a staged approach (myocardial revascularization first followed by PTA) and simultaneous approach (percutaneous coronary intervention immediately followed by PTA at the same time if clinically suitable) are both allowed
   2. the duration from revascularization to PTA should be within 60 days
   3. percutaneous coronary intervention is performed at the time of coronary angiography, using bare metal or drug-eluting stents
3. blood sampling, genotyping, and measurement of biomarkers and microRNA

   a. bood samples (20 mL) are obtained from peripheral arteries in all study subjects before PTA and 10 mL after PTA and are prepared and stored for enzyme-linked immunosorbent assay (ELISA), genotyping and measurement of microRNAs in plasma and peripheral blood mononuclear cells
4. outcome follow-up a. clinical outcomes are obtained by chart review if the patient is still in the hospital and followed up by clinic visit, telephone call or direct contact with participants or subjects' family at 30 days after indexed PTA if the patient has been discharged from the hospital and every 6 months thereafter

ELIGIBILITY:
Inclusion Criteria:

* Known LEAD (documented by previous angiography or sonography performed by the operators) admitted for elective PTA

Exclusion Criteria:

* Known CAD or unstable angina within past 3 months
* Acute myocardial infarction within past 6 months
* Known CAD status posterior percutaneous coronary intervention or bypass surgery within past 6 months
* Planning to do bypass surgery for known LEAD\
* Pregnancy
* Documented active malignancy
* Needing emergency PTA

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to Composite of Major Adverse Cardiac Event (MACE) | up to 48 months
  cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and any unplanned coronary revascularization

SECONDARY OUTCOMES:
MACE between the Screening and 30 days after PTA | 30 days after indexed PTA
  cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and any unplanned coronary revascularization
Time to Composite of major coronary events | Up to 48 months
  fatal or nonfatal myocardial infarction, recurrent angina pectoris, and any unplanned coronary revascularization

OTHER OUTCOMES:
Time to death from any cause | Up to 48 months
  total mortality
Time to congestive heart failure requiring hospitalization | Up to 48 months
  congestive heart failure requiring hospitalization
Time to any coronary revascularization | Up to 48 months
  planned or unplanned coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Hsing Chao, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Background] Chang SH, Tsai YJ, Chou HH, Wu TY, Hsieh CA, Cheng ST, Huang HL. Clinical predictors of long-term outcomes in patients with critical limb ischemia who have undergone endovascular therapy. Angiology. 2014 Apr;65(4):315-22. doi: 10.1177/0003319713515544. Epub 2013 Dec 19. PMID 24357434
- [Background] Monaco M, Stassano P, Di Tommaso L, Pepino P, Giordano A, Pinna GB, Iannelli G, Ambrosio G. Systematic strategy of prophylactic coronary angiography improves long-term outcome after major vascular surgery in medium- to high-risk patients: a prospective, randomized study. J Am Coll Cardiol. 2009 Sep 8;54(11):989-96. doi: 10.1016/j.jacc.2009.05.041. PMID 19729114
- [Background] Duran NE, Duran I, Gurel E, Gunduz S, Gol G, Biteker M, Ozkan M. Coronary artery disease in patients with peripheral artery disease. Heart Lung. 2010 Mar-Apr;39(2):116-20. doi: 10.1016/j.hrtlng.2009.07.004. PMID 20207271
- [Derived] Chen IC, Lee CH, Chao TH, Tseng WK, Lin TH, Chung WJ, Li JK, Huang HL, Liu PY, Chao TK, Chu CY, Lin CC, Hsu PC, Lee WH, Lee PT, Li YH, Tseng SY, Tsai LM, Hwang JJ. Impact of routine coronary catheterization in low extremity artery disease undergoing percutaneous transluminal angioplasty: study protocol for a multi-center randomized controlled trial. Trials. 2016 Feb 29;17(1):112. doi: 10.1186/s13063-016-1237-0. PMID 26927298